CLINICAL TRIAL: NCT02431728
Title: The Effect of Melatonin Upon Post-Acute Withdrawal Among Males in a Residential Treatment Program: A Randomized, Double Blind, Placebo, Controlled Trial
Brief Title: The Effect of Melatonin Upon Post-Acute Withdrawal Among Males in a Residential Treatment Program
Acronym: M-PAWS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duquesne University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DuquesneU
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2015-08

CONDITIONS: Substance Withdrawal Syndrome
Keywords: Melatonin; Post-acute withdrawal symptoms; Anxiety; Depression; Insomnia; Stress; Substance withdrawal syndrome
MeSH Terms: conditions — Substance Withdrawal Syndrome; Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders | interventions — Melatonin; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin (Active Comparator): capsule containing 5mg melatonin plus cellulose
  Interventions: Dietary Supplement: Melatonin
- Matched Placebo (Placebo Comparator): capsule containing cellulose
  Interventions: Dietary Supplement: Matched Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — 5 mg capsule p.o. at bedtime daily
  Other Names: N-acetyl-5-methoxytryptamine
  Arms: Melatonin
Dietary Supplement: Matched Placebo — 5 mg capsule p.o. at bedtime daily
  Other Names: Vegetable fiber
  Arms: Matched Placebo

SUMMARY:
Individuals recovering from drug and/or alcohol addiction initially experience the symptoms of acute withdrawal before experiencing the symptoms of post-acute withdrawal (PAWS). PAWS include a wide array of emotional and psychological symptoms such as anxiety, sleep disturbances, depression, and stress. Previous studies have shown that melatonin therapy was beneficial to alleviate anxiety, depressive symptoms, and sleep disturbances. However, no randomized, double-blind, placebo controlled trials have been conducted in males who are experiencing PAWS. The purpose of this study is to investigate the effect of 5 mg melatonin given nightly for four weeks on weekly assessed, self-reported anxiety, depressive symptoms, insomnia, and stress in males with PAWS who reside in a residential treatment center.

DETAILED DESCRIPTION:
Approval was obtained from the Institutional Review Board at Duquesne University prior to the study implementation. The trial was a single-center, randomized, double-blind, matched placebo-controlled, parallel-group trial conducted in males 18 years of age and older who are in a residential treatment program for chemical dependency at the Salvation Army Harbor Light Center (865 West North Avenue, Pittsburgh, Pennsylvania, 15233) in the United States of America. Convenience sampling was used to recruit individuals from July 2015 to December 2015. A total sample of 70 participants were enrolled and block randomized with an allocation ratio of 1:1 for the interventions. Financial compensation of $5.00 U.S. was initiated at Day 7 and continued at each follow-up (Day 14, Day 21 & Day 28). Intention-to-treat and complete case analyses were conducted. No interim analysis was performed to assess efficacy. Participants completed study materials in a designated room at the center.

Briefly, this study involved the completion of four validated surveys assessing self-reported perceived severity of anxiety (Generalized Anxiety Disorder Scale; GAD-7), depression (Personal Health Questionnaire Depression Scale; PHQ-8), stress (Perceived Stress Scale; PSS-14), sleep complaints and how is sleep affecting daily life (Pittsburgh Sleep Symptom Questionnaire - Insomnia; PSSQ-1) at five time points (Baseline, Day 7, Day 14, Day 21, and Day 28). To address any adverse events relating to the interventions, the participant was encouraged to report any perceived adverse events to the investigator. To protect the anonymity and confidentiality of the participants, all paperwork were de-identified but contained their unique identification number.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 years of age and older who are actively participating in therapy at a residential treatment program
* Willingness to participate in the 4-week study
* Willingness to provide self-reported demographic, social, medical, medication, preventive, and mental health histories
* Willingness to complete self-assessments of anxiety, depression, insomnia, and stress at designated time intervals
* Willingness to administer daily before bed a capsule containing either 5 mg melatonin plus vegetable fiber filler or only the vegetable fiber filler without melatonin (i.e., the matched placebo).
* English speaking

Exclusion Criteria:

* Patients already taking melatonin
* Adverse history with melatonin supplementation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The effect of melatonin or placebo on the change in anxiety as measured by the Generalized Anxiety Disorder (GAD-7) scale | Baseline, Day 7, Day 14, Day 21, Day 28
  The GAD-7 assesses the perceived severity of anxiety through a 7-item scale that assesses anxiety as measured by a symptom checklist over the last two weeks. It employs a four point scale with the response options "Not at all" (0 pts), "Several days" (1 pt), "More than half the days" (2 pts), and "Nearly every day (3 pts). Severity is based on the sum total where 15 - 21 is considered "severe anxiety". The GAD-7 also asks a question about how difficult have these problems contributed to the activities of daily living, responses range from "Not difficult at all" to "Extremely difficult."
The effect of melatonin or placebo on the change in depressive symptoms as measured by the Personal Health Questionnaire Depression Scale (PHQ-8) | Baseline, Day 7, Day 14, Day 21, Day 28
  The PHQ-8 assesses the perceived degree of depression through an 8-item scale that assesses if the individual indicates symptoms over the last two weeks. It employs a four point scale with the response options "Not at all" (0 pts), "Several days" (1 pt), "More than half the days" (2 pts), and "Nearly every day (3 pts). The higher the sum total the greater the degree of depression; for example, a score of ≥20 is considered severe major depression.
The effect of melatonin or placebo on the change in sleep symptoms as measured by the Pittsburgh Sleep Symptom Questionnaire - Insomnia (PSSQ-1) | Baseline, Day 7, Day 14, Day 21, Day 28
  It is a 13-item scale with two subscales: Sleep complaints and How sleep is affecting daily life and assesses their experience during the past month. It employs a six point scale to assess for "Sleep complaints" with response options "Never" (0 pts), "Do not know" (1 pt), "Rarely" (2 pts), "Sometimes" (3 pts), "Frequently" (4 pts) and "Always" (5 pts). It employs a five point scale to assess for "How sleep is affecting daily life," with the response options "Not at all" (0 pts), "A little bit" (1 pt), "Moderately" (2 pts), "Quite a bit (3 pts), and "Extremely" (4 pts). If all criterion questions result in a "Yes," then one can assign a diagnosis of insomnia disorder.
The effect of melatonin or placebo on the change in stress as measured by the Perceived Stress Scale (PSS-14) | Baseline, Day 7, Day 14, Day 21, Day 28
  The PSS-14 assesses the perceived stress through a 14-item scale that asks about the thoughts and feelings of the individual during the past month. It employs a five point scale with the response options "Never" (0 pts), "Almost Never" (1 pt), "Sometimes" (2 pts), "Fairly Often (3 pts), and "Very Often" (4 pts). In scoring the scale, scores are obtained by reversing the scores on items 4, 5, 6, 7, 9, 10, and 13 because these questions are positively stated items. The scores are summed with higher score indicating more perceived stress.

SECONDARY OUTCOMES:
Patient health histories (social, medical, medication, preventive, and mental health) | Baseline
  Patient health histories were used to collect key information that may be used to further identify relevant data that have the potential be used to formulate other studies that the self-reported scales do not assess. Also, the histories were used to measure the effect of confounding and moderating factors.
The number of reported adverse effects | Day 7, Day 14, Day 21, Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Giannetti, Ph.D., Principal Investigator — Duquesne University
Locations (1):
- Salvation Army Harbor Light Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
All data were in aggregrate with no personal identification.